CLINICAL TRIAL: NCT04846855
Title: Regional Anesthesia for Totally Awake Upper Limb Surgery in PEDiatric Population- RAPATED
Brief Title: Regional Anesthesia for Totally Awake Upper Limb Surgery in PEDiatric Population
Acronym: RATAPED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-004504-35
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Anesthesia, Local; Pediatric ALL
Keywords: surgery; local anesthesia; Pediatric; Ropivacaine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: monocentric, interventional, longitudinal, prospective, non-comparative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine 35% (Experimental): Local Anesthesia with Ropivacaine
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: local anaesthetic injection — Realization by the anesthesiologist of the local anesthesia by single dose of ropivacaine 0.35% in perinervous under ultrasound with distraction by a tablette.

SUMMARY:
Peripheral loco-regional anesthesia (LRA) for anesthetic purposes is a technique widely used in adults for upper limb surgery. In pediatrics, LRA is not classically considered on its own. It is usually performed for analgesic purposes during sedation or general anesthesia. It is entirely possible to carry out awakened peripheral blocks in communicating children, of school age, thus avoiding the issues of GA in pediatrics, in particular in an emergency context. The use of Emla anesthetic skin patches for punctures (perfusion and LRA) as well as the viewing of cartoons on touch tablets during treatment can improve the perception of painless care such as LRA and treatment.

In pediatrics, only ropivacaine at a concentration of 0.2% has Marketing Authorization in pediatrics in children under 12 for the production of peripheral blocks. On the basis of the experience of the Claude Galien Private Hospital in this area, it seems interesting to assess the feasibility of upper limb surgery under anesthetic LRA alone with a dose of ropivacaine at the concentration 0.35% in communicating children, of school age.

DETAILED DESCRIPTION:
Peripheral loco-regional anesthesia (LRA) for anesthetic purposes is a technique widely used in adults for upper limb surgery. It allows peripheral surgeries to be performed without putting the patient to sleep and thus avoiding certain disadvantages of general anesthesia (GA).

In pediatrics, LRA is not classically considered on its own. It is usually performed for analgesic purposes during sedation or GA.

Subject to respecting a strict protocol and taking advantage of considerable developments in the field of LRA, it is entirely possible to carry out awakened peripheral blocks in communicating children, of school age, thus avoiding the pitfalls of GA in pediatrics, in particular in an emergency context (inhalation on a full stomach, respiratory risk in children with colds, inhalational anesthesia with an anxiety mask, postoperative vomiting nausea, disorientation and delusions upon waking ...) Indeed, the exclusive use of ultrasound, the use of adapted needles, the improvement of knowledge in sono-anatomy, the reduction in doses and concentrations of local anesthetics are all developments in the field of LRA allowing to improve the conditions of safety, comfort for the patient and success of the technique.

Beyond technical considerations, there are ways to improve the child's experience with care. The use of Emla anesthetic skin patches for punctures (perfusion and ALR) as well as the viewing of cartoons on touch tablets during treatment can improve the perception of painless care such as ALR and treatment. charge in the operating room.

In pediatrics, only ropivacaine at a concentration of 0.2% has Marketing Authorization in pediatrics in children under 12 for the production of peripheral blocks. Higher concentrations of ropivacaine, used in several pediatric studies, have nevertheless shown their good tolerance and their efficacy Under reserve not to exceed 3mg / kg and to use concentrations up to 0.5% On the basis of these arguments, and with the experience of the Claude Galien Private Hospital in this area, it seems interesting to assess the feasibility of upper limb surgery under anesthetic ALR alone with a dose of ropivacaine at the concentration 0.35% in communicating children, of school age.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6 to 12.
* Able to understand and express themselves.
* Intended for orthopedic surgery of the upper limb involving the hand, wrist, forearm or elbow.
* ASA class 1-2.
* Patient who has given free and informed consent.
* Parent present having given their free and informed consent.
* Affiliated patient or beneficiary of a social security scheme

Exclusion Criteria:

* Refusal of the child and / or parent to participate in the study.
* Immediate vital emergency.
* Duration of planned surgery> 1h30.
* History of allergy to LA.
* Contraindication to carrying out ALR (local infection, pathology contraindicating ALR, preoperative neurological deficit).
* Refusal by the surgeon.
* Child already sedated or premedicated in the emergency room.
* Digital tablet not available.
* Patient participating in another clinical study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
LRA success | 2 hours
  percentage of children in whom ALR and surgery were performed without additional sedation or general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Sende, PHD, Principal Investigator — Ramsay santé
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided